CLINICAL TRIAL: NCT01983150
Title: Effect of a Smartphone Intervention on Quitting Smoking in a Young Adult Population of Smokers: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial to Test the Effect of a Smartphone Quit Smoking Intervention on Young Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19275
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Cigarette Smoking
Keywords: Population Health; Smoking cessation; Young adults; Cancer prevention; Tobacco control strategies; Behaviour modification; Social Media; Smartphone technology
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Media Exposure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crush the Crave Application (Experimental): Crush the Crave (CTC) intervention group will receive a quit smoking smartphone intervention via the internet that is based on scientific findings related to tobacco use among young adults. It is a multi-component intervention informed by evidence on quitting smoking. The app was developed with the input of key experts in the field of smoking cessation, was assessed against Fiore's practice guidelines for treating tobacco use and dependence, and was tested with eight focus groups of male and female young adult smokers (n=57) on functionality, look and feel and usability, as well as being piloted by over 300 smokers.
  Interventions: Behavioral: Crush the Crave Application
- On the Road to Quitting - Self Help (Active Comparator): The control group will receive an evidence-based self-help guide known as "On the Road to Quitting"(45) that has been developed by Health Canada for young adult smokers. Participants will be able to both view the self-help guide via the internet and will receive a printed version of the guide.
  Interventions: Behavioral: On the Road to Quitting - Self Help

INTERVENTIONS:
Behavioral: Crush the Crave Application — Crush the Crave (CTC) allows users to customize a quit plan by choosing a quit date and then deciding whether to quit now or cut down the number of cigarettes they smoke every week up to the quit date. CTC reminds users of money saved and health improvements. Based on contingency reinforcement, rewards are provided, which smokers can then choose to share with their social network via Facebook. Supportive text messages tailored to their specific quit plan and where they are in the quitting experience are provided. CTC allows tracking of daily smoking habits and cravings as well as craving triggers or psychosocial determinants by recording when, where and why smoking occurred. Online distractions to help smokers deal with cravings are provided.
  Other Names: Android; iPhone; Mobile phone; Behavior change; Quit smoking; Social media; Facebook
  Arms: Crush the Crave Application
Behavioral: On the Road to Quitting - Self Help — The control group will receive an evidence-based self-help guide known as "On the Road to Quitting" that has been developed by Health Canada for young adult smokers. Participants will be able to both view the self-help guide via the internet and will receive a printed version of the guide.
  Arms: On the Road to Quitting - Self Help

SUMMARY:
The primary aim of this study will be to determine the effectiveness of a smartphone delivered app for young adult smokers on quitting smoking.

DETAILED DESCRIPTION:
The principle study purpose of the randomized controlled trial is to determine the effectiveness of a smartphone delivered app for young adult smokers on smoking cessation at six months using a randomized controlled trial. Secondary aims of this study include examining: 1) proximal outcome measures of cessation behaviour; 2) satisfaction, extent of app use and use of NRT and other cessation services; 3) mediators of cessation outcomes between conditions; and 4) the incremental cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 29 years
* Currently smoking cigarettes daily or occasionally
* Residing in Canada
* Considering quitting smoking in the next 30 days
* Have an Android or iPhone OS smartphone
* Able to provide informed consent
* English comprehension
* Not referred by a study participant

Exclusion Criteria:

- opposite of the above

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1601 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
30 day point prevalence of abstinence | 6 months
  30 day point prevalence of abstinence at 6 months,operationalized as not having smoked any cigarettes, even a puff, or used other tobacco in the last 30 days.

SECONDARY OUTCOMES:
7-day abstinence | 6 months
  7 day point prevalence of abstinence at 6 months,operationalized as not having smoked any cigarettes, even a puff, or used other tobacco in the last 30 days
Number of quit attempts | 6 months
  How many times did you stop using tobacco for 24 hours or longer over the past six months?
Consumption of cigarettes | Baseline and at 6 months
  Reduction in the consumption of cigarettes since baseline and behavioural intentions to quit smoking using questions from the Minimal Dataset and nicotine withdrawal using the Fagerstrom test for nicotine dependence.
Satisfaction and App Utilization | 6 months
  Satisfaction with program, app utilization metrics, and use of smoking cessation services (NRT, health professional consults,medications and quitline counseling)
Psychosocial measures | Baseline and at 6 months
  Beliefs, attitudes and social norms using the Smoking Attitudes Scale, stress using the 14-item Perceived Stress Scale, self-efficacy using Etter's 12 items, and perceived social support using the modified 7-item subjective support subscale of the Duke Social Support Index.

CONTACTS AND LOCATIONS:
Overall Officials: Neill B Baskerville, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Baskerville NB, Struik LL, Guindon GE, Norman CD, Whittaker R, Burns C, Hammond D, Dash D, Brown KS. Effect of a Mobile Phone Intervention on Quitting Smoking in a Young Adult Population of Smokers: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Oct 23;6(10):e10893. doi: 10.2196/10893. PMID 30355563
- [Derived] Baskerville NB, Struik LL, Dash D. Crush the Crave: Development and Formative Evaluation of a Smartphone App for Smoking Cessation. JMIR Mhealth Uhealth. 2018 Mar 2;6(3):e52. doi: 10.2196/mhealth.9011. PMID 29500157
- [Derived] Baskerville NB, Struik LL, Hammond D, Guindon GE, Norman CD, Whittaker R, Burns CM, Grindrod KA, Brown KS. Effect of a mobile phone intervention on quitting smoking in a young adult population of smokers: randomized controlled trial study protocol. JMIR Res Protoc. 2015 Jan 19;4(1):e10. doi: 10.2196/resprot.3823. PMID 25599695